CLINICAL TRIAL: NCT07034729
Title: Effect of Emotıonal Intellıgence Skılls Development Traınıng on Nurses' Fear of Intımacy and Care Behavıors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Başakşehir Çam & Sakura City Hospital (Other Government)
Responsible Party: Principal Investigator, Demet Duman, Nursing manager, Başakşehir Çam & Sakura City Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2022-321
Record Dates: First submitted 2025-05-24; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2024-05

CONDITIONS: Emotional Intelligence; Care Eliciting Behavior
Keywords: care behaviors; fear of ıntimacy; emotional intelligence

STUDY DESIGN:
Intervention Model Description: The research was designed as a single-center, experimental study based on a randomized control group pre-test-post-test design.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): The scale was applied to the intervention group.By creating the Emotional Intelligence Skills Development Training Module, participants in the initiative group will be trained in 6 modules.
  Interventions: Behavioral: training to develop emotional intelligence skills
- non-intervention (No Intervention): Only the scale was applied to the non-intervention group.

INTERVENTIONS:
Behavioral: training to develop emotional intelligence skills — 2 hours in a week, 6 week training
  Arms: intervention group

SUMMARY:
Emotional intelligence is a type of intelligence that can be developed, which gives individuals the ability to understand and express emotions to the other party. Studies have shown that individuals with a developed level of emotional intelligence can analyze their own and others' emotions and thoughts well, manage their emotions, interact positively with their environment, and are successful in interpersonal relationships and professional skills. Intimacy, on the other hand, is the ability to truly share the true self with another person. When fear develops regarding the concept of intimacy, which affects interpersonal relationships; individuals' healthy communication with other individuals is restricted, and feelings and behaviors that avoid intimacy may occur. The concept of "care" in nursing is related to the relationship between the nurse and the healthy/patient individual and the care process.

In this study, it was planned to examine the effect of fear of intimacy and care behaviors of nurses by providing emotional intelligence skills development training to nurses in line with literature data. The research was designed as a single-center, randomized control group pretest-posttest experimental study.

DETAILED DESCRIPTION:
The research sample consisted of bachelor's degree nurses who were working at Başakşehir Çam and Sakura City Hospital- Neurology Orthopedics Hospital between November 2023 and May 2024 and who agreed to participate in the study and had at least one year of work experience [98 intervention group - 98 control group]. The intervention and control groups were determined using a random numbers table from the simple random sampling method. In line with Daniel Goleman's Emotional Intelligence Model, the Emotional Intelligence Skills Development Training Module was created and the participants in the intervention group were trained in 6 modules. Before the first module of the training was implemented, the Nurse Information Form prepared via Google Forms, the Revised Schutte Emotional Intelligence Scale, the Fear of Intimacy Scale, and the Care Behaviors-24 Scale were filled out. When the 6th Module of the training was completed, the Revised Schutte Emotional Intelligence Scale, the Fear of Intimacy Scale, and the Care Behaviors-24 Scale were filled out. The participants in the control group of the study were asked to fill out the Nurse Information Form, Revised Schutte Emotional Intelligence Scale, Fear of Intimacy Scale and Caring Behaviors-24 Scale prepared via Google Forms simultaneously with the first module. No intervention was applied to the control group. At the end of Module 6 of the training, the Revised Schutte Emotional Intelligence Scale, Fear of Intimacy Scale and Caring Behaviors-24 Scale were filled out simultaneously with the intervention group. The scales were re-applied to the intervention and control groups 3 months later. Emotional intelligence skills training was given and its effects on fear of intimacy and caring behaviors were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Actively taking part in the care of a healthy/sick individual for at least 1 year
* Having a bachelor's degree in nursing
* Being willing to participate in the study

Exclusion Criteria:

* Not being in the initiative group and not having attended more than 2 sessions of training
* Leaving the study voluntarily

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2023-11-12 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Revised Schutte Emotional Intelligence Scale | Evaluation was made at the beginning of the 1st week of training and at the end of the 6th week of training.
  Participants' emotional intelligence skills will be evaluated before and after the training using a scale. The scale consists of 41 questions and is evaluated with a 5-point Likert-type scale.
  The total score in the Revised Schutte Emotional Intelligence Scale, adapted to Turkish in the 2011 study by Tatar, Tok and Saltukoğlu, indicates the level of emotional intelligence. Scores between 41 and 90 indicate low emotional intelligence, scores between 91 and 150 indicate medium emotional intelligence, and scores between 151 and 205 indicate high emotional intelligence. As the score increases, the level of emotional intelligence increases.

SECONDARY OUTCOMES:
Fear of Intimacy Scale | It was evaluated at the beginning of the 1st week of training and at the end of the 6th week of training.
  Pre- and post-training evaluations were made using the fear of intimacy scale. The scale consists of 35 questions and is evaluated with a 5-point Likert-type scale.The minimum score on the scale is 35 and the maximum score is 175. It is accepted that the fear of intimacy will increase as the score on the scale increases.
Caring Behaviors-24 Scale | Evaluated before the 1st week of training and at the end of the 6th week of training
  The Care Behaviors-24 Scale was used for pre- and post-training evaluations. The scale consists of 24 questions and is evaluated with a 6-point Likert-type scale.
  A minimum of 24 and a maximum of 144 points can be obtained from the research. It is accepted that as the score obtained increases, care behaviors improve.

CONTACTS AND LOCATIONS:
Locations (1):
- Basaksehir Cam and Sakura Cıty Hospıtal, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Because the study was not published

REFERENCES:
- [Background] Erkayıran O. (2016). The Effect of Emotional Intelligence Skills Development Training on Interpersonal Relations of Nursing Students, Adnan Menderes University Health Sciences Institute Master Thesis, 2016, Aydın.